CLINICAL TRIAL: NCT04907604
Title: European platforM to PromOte Wellbeing and HEalth in the woRkplace
Brief Title: European platforM to PromOte Wellbeing and HEalth in the Workplace (EMPOWER)
Acronym: EMPOWER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Universidad Autonoma de Madrid (Other); Erasmus University Rotterdam (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); University of York (Other); Fondazione Adapt (Unknown); Schweizer Paraplegiker Forschung (Other); Australian National University (Other); City of Turku (Other Government); Ómada Interactiva SLL (Unknown); Instytut Medycyny Pracy Imienia Prof. Dra Med. Jerzego Nofera W Lodzi (Unknown); University of Lodz (Unknown); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PIC-39-20; Grant Agreement:848180 (Other Grant/Funding Number: Research and Innovation Framework Programme SC1-BHC-22-2019)
Record Dates: First submitted 2021-04-28; First posted 2021-06-01 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Stress; Anxiety; Depression; Insomnia
Keywords: Mental health; Well-being; Workplace
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: It will conduct a stepped wedge cluster randomized trial with randomization on the company level, each company representing one cluster. The design involves random and sequential crossover of clusters from control to intervention until all clusters are exposed. Data collection continues throughout the study so that each cluster contributes observations under both control and intervention observation periods. This design was selected in order to retain the power of randomization while offering all companies enrolled in the trial the desirable intervention.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First intervention group (Other): Clusters 1 and 2 (group 1) will start the intervention at month 1, immediately after completing the baseline assessment. After 7 weeks of using the app and having access to the EMPOWER website (with material related to the anti-stigma campaign and recommendations for employees to deal with psychosocial risk factors), they will answer a post-treatment assessment protocol through the app.
  Interventions: Device: A multi-modal and integrative e-health platform aimed at promoting health and reducing the negative impact of mental problems in the workplace
- Second intervention group (Other): Clusters 3 and 4 (group 2) that serve as control group of cluster 1 and 2 (group 1), will also complete the assessment at T1. Clusters 3 and 4 (group 2) will start the intervention in step 2, after completing the second assessment.
  Interventions: Device: A multi-modal and integrative e-health platform aimed at promoting health and reducing the negative impact of mental problems in the workplace
- Third intervention group (Other): Clusters 5 and 6 (group 3), that serve as control group of group 1 and 2, will also complete the assessment at T2. Clusters 5 and 6 (group 3) will start the intervention in step 3. All clusters will answer a total of five assessments
  Interventions: Device: A multi-modal and integrative e-health platform aimed at promoting health and reducing the negative impact of mental problems in the workplace

INTERVENTIONS:
Device: A multi-modal and integrative e-health platform aimed at promoting health and reducing the negative impact of mental problems in the workplace — It addresses six main domains: improving awareness of mental health problems and reducing stigma; reducing psychosocial risk factors in the workplace; improving wellbeing and reducing psychological symptoms; ensuring early detection of mental disorders; promoting healthy behaviours and lifestyles; and facilitating early return to work.

SUMMARY:
EMPOWER is a multidisciplinary research and innovation effort aiming to developing, implementing, evaluating and disseminating the effectiveness and cost-effectiveness of a modular eHealth intervention platform to promote health and well-being, reduce psychological distress, prevent common mental health problems and reduce their impact in the workplace. In collaboration with stakeholders, we will adapt existing effective interventions focused on different components (awareness and stigma, workplace conditions and psychosocial factors, stress, common mental health symptoms, early detection, comorbidity, lifestyle, and return to work) to created a combined online modular platform feasible in various workplace settings by culturally and contextually adapting it. The intervention will be implemented through a stepped wedge cluster randomized trial directed to employees and employers of small and medium sized enterprises and public agencies from three European countries (Spain, Finland and Poland) and United Kingdom. Both qualitative and quantitative methods will be used in the evaluation of the individual health outcomes, cost-effectiveness (from a social, economical, employer and employees perspective), and implementation facilitators and barriers. Implementation strategies relevant to the uptake of the EMPOWER intervention will be identified, including a realistic appraisal of barriers to uptake as well as evidence-based solutions to these barriers. Through scaling-up pre-existing effective and cost-effective interventions, EMPOWER is aimed at addressing the overarching challenges from different perspectives, including individual level (e.g., addressing stigma, mental health, well-being and lifestyles, taking into account legal, cultural and gender issues) and organizational level. The main outcomes effort will help employees, employers and policymakers in decision processes of new legal and contractual framework at EU and national level covering the new economy landscape.

DETAILED DESCRIPTION:
The EMPOWER Project's main objective is to develop, test and evaluate a multi-modal and inclusive e-Health platform, compiling the most feasible, brief and cost-effective interventions currently available in Europe to promote health and wellbeing, prevent mental health problems and reduce the impact of mental health problems in the workplace.

Specifically, three intervention levels will be represented by interventions within the eHealth platform that are specially designed for the relevant populations and desired outcomes:

1. Universal (primary) prevention: interventions to improve awareness and reduce stigma; to reduce psychosocial risk factors and providing early detection of mental disorders.
2. Secondary prevention programs: interventions designed to improve wellbeing and reduce psychological distress and to promote healthy lifestyles. EMPOWER individual eHealth intervention will be based on the following components:

   * Psychoeducational material.
   * Challenges
   * Tracking
3. Tertiary prevention program: return to work intervention. The intensive collaborative approach will design strategies to overcome the barriers that have already been identified for the widespread implementation of programs to promote wellbeing and reduce mental health problems in the workplace. EMPOWER aims to address the increasing burden of mental health problems in the workplace and improve mental health in the EU working population, having a positive impact on productivity. Partners from the consortium are coming from countries such as Spain, Italy, Netherlands, Poland, UK, Switzerland and Australia.

An eHealth platform to reduce the impact of mental health problems at the workplace Mental health problems cause an enormous burden both for the individual and the society. A number of interventions have been developed to promote wellbeing and prevent or treat mental disorders in the workplace. Attempts to implement interventions by means of digital technologies have had statistically significant but minimally positive effects in reducing overall mental health problems, such as depression, anxiety and stress. However, most eHealth interventions focus on a single mental health condition and neglect comorbidity, particularly in the case of the more common mental disorders. Although effective and cost-effective workplace interventions are available, widespread implementation face a number of barriers. The stigma and discrimination at the workplace have been associated with delayed access to treatment, weakened social support, difficulties in the performance of occupational and social roles, unemployment, and diminished self-esteem. Although anti-stigma interventions targeting the general population and workplace settings have been implemented, there is room for improvement.

Collaboration among stakeholders is essential when developing and implementing effective interventions to reduce the impact of mental health problems at the workplace and evaluate their impact. The organization of work is rapidly changing. This growing diversity of what it means to work makes it clear that addressing mental health issues at the workplace will require ingenuity and flexibility to tailor interventions to the realities of the workplace setting.

The Framework Directive on Occupational Safety and Health, 89/391/EEC, lays down the employers' general duty to ensure workers' health and safety, "addressing all types of risk". Although the Framework does not explicitly address mental health issues in the workplace, it implicitly addresses them since it requires the employer to be aware of and address all types of health-related risks. At the same time, the European Commission's 2008 European Pact for Mental Health and Well-being20 and the 2016 European Framework for Action on Mental Health and Well-being21 have clearly raised the issue of mental health as a public health priority across society and the economy, mentioning workplace mental health as one target area. Although there has not as yet been a direct regulatory focus on mental health in the workplace, there is certainly a general consensus that it is incumbent on European employers to adequately identify and address known psychosocial risks.

Due to the fragmented landscape of interventions and related implementation barriers, there is an urgent need for a multi-modal and integrative eHealth platform aimed at reducing mental health problems in the workplace and improving employees' wellbeing, by compiling the most feasible, brief and cost-effective interventions currently available in Europe. The platform will take advantage of proven cost-effective tools and address the need to reduce stigma, increase help-seeking behaviour, raise awareness about and minimalize psychosocial risks, improve self-management strategies, taking into account mental and physical comorbidities, and promote a healthy lifestyle - all while considering gender and cultural differences that impact successful implementation. This is especially relevant for small and medium enterprises (SMEs), which represent the majority of all enterprises in the EU but have very limited resources. The development and implementation of a multi-modal and integrative eHealth platform should, finally, be guided and supported by close collaboration with stakeholders, including employee and employer organisations, insurance companies, patient associations, and health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Having a mobile phone with internet access
* Having sufficient knowledge of the local language
* Accepting the informed consent.
* Being employed at the time of recruitment (baseline)

Exclusion Criteria:

* Younger than 18
* Not having sufficient knowledge of the local language
* Being unemployed at the time of recruitment (baseline)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 729 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | at both 7 weeks and 3-month follow-up
  Change in depressive symptomatology for employees, measured with the Patient Health Questionnaire-9 (PHQ-9) sum score. It ranges from 0 to 27, with higher scores indicating more severe symptomatology. A score higher than 19 is considered as indicative of high risk of depression

SECONDARY OUTCOMES:
Anxiety symptoms | at both 7 weeks and 3-month follow-up
  Change in anxiety symptoms (by means of the Generalized Anxiety Disorder-7-GAD-7- total scores). The total score ranges from 0 to 21, with higher scores indicating higher level of anxiety.
Perceived stress | at both 7 weeks and 3-month follow-up
  Change of perceived stress measured with the Perceived Stress Scale-4 (PSS-4). The total score ranges from 0 to 16, with higher scores correlating with higher levels of stress.
Insomnia severity | at both 7 weeks and 3-month follow-up
  Change in insomnia severity uisng three items of Insomnia Severity Index (ISI). We will calculate a total score which will range from 0 to 16. Higher scores will indicate severe levels of insomnia.
Well-being | at both 7 weeks and 3-month follow-up
  Change in well-being (assessed with the World Health Organization-5; WHO-5 scale). The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Olaya, Principal Investigator — Parc Sanitari Sant Joan de Déu

IPD SHARING:
Plan to Share IPD: No
Despite a plan to make IPD available is not being decided yet, the aim of EMPOWER is to follow the FAIR criteria for research data. The data produced and/or used in the project should be assessable for and intelligible to third parties in contexts such as scientific scrutiny and peer review (e.g. data are provided in a way that judgments can be made about their reliability and the competence of those who created them). In that regard, EMPOWER has the intention to make (part of) the research data Findable, Accessible, Interoperable and Re-usable (FAIR).

REFERENCES:
- [Derived] Salvador-Carulla L, Lukersmith S, Woods CE, Chen T, de Miquel C. A protocol using mixed methods for the impact analysis of the implementation of the EMPOWER project: an eHealth intervention to promote mental health and well-being in European workplaces. BMJ Open. 2025 Apr 9;15(4):e082219. doi: 10.1136/bmjopen-2023-082219. PMID 40204313
- See also: EMPOWER project webpage — http://empower-project.eu/